CLINICAL TRIAL: NCT02850601
Title: Dexamethasone Solution and Dexamethasone in Mucolox™ for the Treatment of Oral Lichen Planus
Brief Title: Dexamethasone Solution for the Treatment of Oral Lichen Planus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Herve Y. Sroussi, D.M.D.,Ph.D., Oral Medicine Attending, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016D003018
Record Dates: First submitted 2016-07-26; First posted 2016-08-01 (Estimated); Results first posted 2021-05-14 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-05

CONDITIONS: Lichen Planus
Keywords: Oral lichen planus; Dexamethasone solution
MeSH Terms: conditions — Lichen Planus; Lichen Planus, Oral | interventions — Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dexamethasone solution (Experimental): Dexamethasone 0.5 mg/mL, 5ml TID for 4 weeks
  Interventions: Drug: Dexamethasone
- Dexamethasone solution in Mucolox™ (Active Comparator): Compounded dexamethasone 0.5 mg/mL in Mucolox™, 5ml TID for 4 weeks
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — Dexamethasone solution 0.5 mg/mL, rinse for 5 minutes and expectorate
  Other Names: Decadron Elixir

SUMMARY:
The objective of this single center, 4-week, open label randomized, phase II study is to evaluate and characterize the tolerability and clinical effectiveness of dexamethasone 0.5mg/5ml solution in a mucoadhesive vehicle (Mucolox™) for the treatment of oral lichen planus.

DETAILED DESCRIPTION:
Potentially eligible subjects will be screened by one of the investigators by asking patients to rate their worst oral pain or pain score (0-10) over the previous week (see Appendix). Those answering with at least a score of "7" (1/10) and that meet all other eligibility requirements (see Section 3) will be eligible for enrollment. All patients will sign informed consent for study participation. Each study visit is anticipated to take approximately 45 minutes.

Treatment will be administered on an outpatient basis. Study medication will be prescribed by authorized study staff physicians at no expense for the patient.

Subjects will be evaluated clinically at baseline before starting treatment and at the end of the four-week period, for a total of two visits. Comprehensive subjective and objective data will be collected and intraoral photographs will be obtained. Oral mucosal disease will be evaluated using both patient reported (questions/visual analog scales) and clinician assessed measures.

Subjects will be prescribed compound dexamethasone 0.5mg/5ml solution in Mucolox™ (ARM A) or dexamethasone 0.5mg/5ml solution only (ARM B). All subjects will also receive a prescription for fluconazole 200 mg tablets once-a-week as prophylactic antifungal therapy. Any subjects that are already taking an antifungal oral medication at the time of the study enrollment will continue their prescribed medication and will not need to take the additional weekly fluconazole dose. Subjects will return for evaluation after four weeks at which time the study end-points will be assessed.

If there is worsening of oral lichen planus that requires initiation of new immunomodulatory medications (systemic or topical), patients will remain on treatment, but will be regarded as unevaluable for the primary endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older.
* Patients with symptomatic oral lichen planus (worst VAS sensitivity score ≥ 7 over the last week).

Exclusion Criteria:

* Patients already on topical or systemic steroids.
* Inability to comply with study instructions.
* Uncontrolled intercurrent illness or psychiatric illness/social situations that would limit compliance with study requirements.
* VAS sensitivity score < 7.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-02-07 (Actual); Primary Completion 2019-12-19 (Actual); Study Completion 2019-12-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dexamethasone Solution | Dexamethasone Solution in Mucolox™
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexamethasone Solution | Dexamethasone Solution in Mucolox™ | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Full Range); unit: years] | 80.2 [74 to 84] | 58.8 [45 to 80] | 69.5 [45 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 9 | 21
  Male | 0 | 3 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 12 | 12 | 24
Sensitivity at baseline on a 0-10 scale [Mean (Full Range); unit: units on a scale] — Subjects scored their worse sensitivity while eating over the past week on an 11 point scale (visual analogue scale 0-10). O signifies no sensitivity; 10 maximum sensitivity.
  units on a scale | 8 [7 to 10] | 8 [7 to 10] | 8 [7 to 10]

OUTCOME MEASURES:

1. Primary Outcome: Change in Oral Sensitivity
Description: Subjects scored their worse sensitivity while eating over the past week. This score is substracted from their initial reported sensitivity at baseline.
  Reduction in oral symptoms of the worst sensitivity experienced in the past week on an 11 point scale (visual analogue scale 0-10). O signifies no sensitivity; 10 maximum sensitivity substracted from the same score collected at baseline before the treatment was initiated.
Time Frame: 4 weeks after the start of the trial
Measure: Median (Standard Error); unit: score on a scale
Groups:
- Dexamethasone Rinses: 12 subjects A four-week supply of dexamethasone solution (0.1mg/ml) was dispensed and subjects were instructed to swish for 5 minutes and expectorate with 5 mL of solution, three times a day, and to avoid eating or drinking for 15 minutes
- Dexamethasone in Mucolox Rinses: 12 subjects A four-week supply of dexamethasone in Mucolox at 0.1mg/ml was dispensed and subjects were instructed to swish for 5 minutes and expectorate with 5 mL of solution, three times a day, and to avoid eating or drinking for 15 minutes
Arm/Group | Dexamethasone Rinses | Dexamethasone in Mucolox Rinses
Number analyzed (Participants) | 12 | 12
score on a scale | -4.5 (2.5) | -6.0 (1.5)

ADVERSE EVENTS:
Time Frame: Onset of symptoms were reported 4-5 days after initiating the treatment and lasted 24h. The treatment was interrupted for 2 days and resumed thereafter with no recurrence or any other adverse event. The subject was monitored through study completion (4 weeks after baseline).
Description: Abdominal discomfort 4-5 days after initiating study drug. Study drug was discontinued and event ended 2 days later and did not recur.
Arm/Group | Dexamethasone Solution | Dexamethasone Solution in Mucolox™
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 1/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dexamethasone Solution (N=12) | Dexamethasone Solution in Mucolox™ (N=12)
constipation; abdomional discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) — Stopped study meds and recovered after 1 day

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-21): https://cdn.clinicaltrials.gov/large-docs/01/NCT02850601/Prot_SAP_001.pdf